CLINICAL TRIAL: NCT02205970
Title: Methodological Proposal of Application of Electrical Neurostimulation Transcutaneous (Comparative Study Between Proposed Method of Application Versus Traditional Method in Patients With Primary Dysmenorrhea).
Brief Title: Application of Electrical Neurostimulation Transcutaneous in Patients With Primary Dysmenorrhea.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Fabio Mendes Camilo, Methodological Proposal of Application of Electrical Neurostimulation Transcutaneous (Comparative Study between Proposed Method of Application Versus Traditional method in patients with Primary Dysmenorrhea)., Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFSaoCarlos0001/14; 036/2010 (Other: CEP-FISA/FUNEC)
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Primary Dysmenorrhea
Keywords: TENS; Dysmenorrhea; analgesia; interactive
MeSH Terms: conditions — Dysmenorrhea; Agnosia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: one arm study
Oversight: Data Monitoring Committee: No

ARMS (2):
- TENS active (Active Comparator): TENS (interactive): frequency (90 and 150 pps) and pulse duration (300 and 400μs)
  Interventions: Device: TENS
- TENS sham (Sham Comparator): Placebo lasting 35 minutes.
  Interventions: Device: TENS (sham)

INTERVENTIONS:
Device: TENS — In the active group there was only one application with interactive TENS (n = 42) with the final parameters of frequency between 90 and 150pps and pulse duration between 300 and 400μs and intensity level of tolerance, lasting 35 minutes.
  Other Names: TENS - eletric pulse generator
  Arms: TENS active
Device: TENS (sham) — In the placebo group, there was a simulated single application, following the same procedures as the active TENS group, also for 35 minutes.
  Arms: TENS sham

SUMMARY:
The present study aims to verify the analgesic potential of a new methodological proposal for application for transcutaneous electrical nerve stimulation (TENS interactive) using patients with primary dysmenorrhoea and compare it with placebo in a randomized double blind study with convenience sample.

DETAILED DESCRIPTION:
The denouement will be the intensity of pain from visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* Primary dysmenorrhoea
* Moderate to severe pain

Exclusion Criteria:

* Secondary dysmenorrhea
* Users of intrauterine device
* Cognitive impairment
* Failure to appear for treatment
* Pacemaker use
* Illicit drug use
* Epilepsy
* Skin problems
* Use of pain medication before the application of TENS

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2010-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
measure the pain threshold, used to Visual Analogue Scale (VAS)before and after application | participants will be monitored for 24 hours
  To assess pain intensity, will be used to Visual Analogue Scale (VAS), Assessments with EVA are performed before and after treatment of interactive TENS (proposed method). All selected volunteers were subjected to an application of TENS (active or sham) in a single menstrual cycle.

SECONDARY OUTCOMES:
duration of analgesia after application | 1 week
  check the duration of analgesia after application of interactive TENS (proposed method)

CONTACTS AND LOCATIONS:
Overall Officials: Fábio M. Camilo, teacher, Principal Investigator — Fundação de Educação e Cultura de Santa Fé do Sul